CLINICAL TRIAL: NCT03394248
Title: The Effects of Subconcussive Events on Cognition
Status: Completed | Type: Observational
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Matthew Heller, Assistant Professor, Family Medicine, New York Institute of Technology
Other Study IDs: BHS-1304
Record Dates: First submitted 2017-12-20; First posted 2018-01-09 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Injury
Keywords: Subconcussive head injury
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Vector Mouthguard — The mouthguard will be used by athletes to measure the magnitude and number of impacts throughout one season.

SUMMARY:
The purpose of this study is to determine early detection of concussion for those at risk of developing symptoms and to be able to detect subconcussive cerebral impairment, and thus gaining a better understanding of the injury patterns for concussions in Men's and Women's Collegiate sports.

DETAILED DESCRIPTION:
Description of the Research Subjects will be members of NYIT's Collegiate Athletic Teams. Potential subjects will be informed about the proposed study and asked if the athlete is interested in participating. If the athlete agrees, the key investigator will review the study procedures, what is expected of the subject, and complete the informed consent process. Participation will be completely voluntary and will have no impact on the quality of care the subject will receive. Inclusion and exclusion criteria will then be evaluated by the key investigator to determine if the subject is qualified to participate in this study. Following consent and review of inclusion and exclusion criteria, the subject will be assigned a subject identification number in which is intended to maintain confidentiality of the subject's personal health information. The number will be used for the duration of the study and in all analyses. Once enrolled, the subjects will complete a baseline questionnaire* that will include demographic information and personal history, as well as consent for de-identified information to be shared with a third party, Quadrant Biosciences, for research purposes. The subjects will be evaluated by a series of measurements, ClearEdge, Quadrant Bioscience Salivary Testing, King Devick, and Im PACT, in the preseason, midseason, and postseason, or if they are suspected of a concussion by the athletic trainer or team physician. Visit 1: Baseline Data Collection

* Assessment Tools
* Demographic/Baseline questionnaire*
* ImPACT
* King-Devick
* ClearEdge New York Institute of Technology Institutional Review Board Approved From 07/18/20 to 07/17/21
* Quadrant Bioscience Salivary Testing
* Quadrant Bioscience Salivary Testing Questionnaire
* Estimated Time: 1.5 hours Visit 2: Mid-Season Collection
* Assessment Tools
* ImPACT
* King-Devick
* ClearEdge
* Quadrant Bioscience Salivary Testing
* Quadrant Bioscience Salivary Testing Questionnaire
* Estimated time: 1 hour Visit 3: Post-season Data Collection
* Assessment Tools
* ImPACT
* King-Devick
* ClearEdge
* Quadrant Bioscience Salivary Testing
* Quadrant Bioscience Salivary Testing Questionnaire
* Estimated time: 1 hr Visit 4: If athlete is suspected to have sustained a concussion by the athletic trainer or team physician, the athlete will come for an additional visit
* Assessment Tools
* ImPACT
* King-Devick
* ClearEdge
* Quadrant Bioscience Salivary Testing
* Quadrant Bioscience Salivary Testing Questionnaire
* Estimated time: 1 hr

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years age and younger than 50 years of age
* Subject experiences at least 8Gs of force on at least one occasion, as measured by accelerometer

Exclusion Criteria:

* The subject suffered from any of the following at the time of event leading to a concussion:

  * Loss of consciousness >2 minutes in the field as reported by witness
  * Seizures
  * Intractable vomiting
  * Paralysis
* The subject has been diagnosed with an underlying neurodegenerative condition that may confound test results (e.g. Parkinson's Disease, Alzheimer's Disease)
* The subject has a current or previous spinal cord injury
* The subject is unable to complete assessment tools
* The subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will be members of the NYIT Athletic Teams.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Changes in cognition secondary to impact | 5 months
  A mouthguard with built in sensors to collect data above the predetermined acceleration thresholds. The predetermined threshold for acceleration will be set to 5G in order to collect more data about subconcussive impacts, in addition to concussive impacts

SECONDARY OUTCOMES:
ImPACT Testing | 5 months
  Tool to help detect and assess the severity of concussion in athletes by establishing a baseline of memory and cognitive function
King-Devick Test | 5 months
  Objectively measures visual tracking and saccadic eye movements
C3 Logix | 5 months
  Concussion Assessment application with the ability to track a patient's dynamic vision reflexes and ability to focus on moving objects

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Heller, D.O, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
May share with osteopathic medical research students